CLINICAL TRIAL: NCT06929364
Title: The Role of Probiotics in the Treatment of Endometriosis (ProMetrioS): a Randomised Double-blinded Placebo-controlled Cross-over Trial
Acronym: ProMetrioS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The Gut Microbiome Center (Centar za crijevni mikrobiom) (Other)
Collaborators: Clinical Hospital Centre Zagreb (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: ProMetrioS2024
Record Dates: First submitted 2024-09-17; First posted 2025-04-16 (Actual); Last update posted 2025-04-16 (Actual); Status verified 2025-04

CONDITIONS: Endometriosis; Probiotics
Keywords: endometriosis; probiotics; microbiome
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: I got error for writing 2 arms and that participants and investigator are masked so I had to adapt it.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patient group 1 (Experimental): Arm 1: Probiotic-Placebo Sequence Description: Participants will consume Omni Biotic Stress (multistrain probiotic formulation) once daily for 8 weeks during the first phase, followed by an 8-week washout period, and then placebo once daily for 8 weeks during the second phase.
  Interventions:
  Dietary Supplement: Omni Biotic Stress; Other: Placebo
  Interventions: Dietary Supplement: Omni Biotic Stress; Other: Placebo
- patient group 2 (Experimental): Arm 2: Placebo-Probiotic Sequence Description: Participants will consume placebo once daily for 8 weeks during the first phase, followed by an 8-week washout period, and then Omni Biotic Stress once daily for 8 weeks during the second phase.
  Interventions:
  Other: Placebo; Dietary Supplement: Omni Biotic Stress
  Participants will record adherence and any potential side effects in an online form. Researchers will check the number of used sachets to ensure accuracy of adherence data.
  Interventions: Dietary Supplement: Omni Biotic Stress; Other: Placebo

INTERVENTIONS:
Dietary Supplement: Omni Biotic Stress — Multistrain probiotic formulation (Omni Biotic Stress), 1 sachet daily for 8 weeks
Other: Placebo — Inert powder identical in appearance and taste to probiotic, 1 sachet daily for 8 weeks

SUMMARY:
ProMetrioS is a randomised blinded placebo-controlled cross-over trial investigating the effect of specific multistrain probiotics in patients with endometriosis. The aim of this clinical trial is to determine whether probiotic treatment can significantly modulate gut microbiome composition and functionality in endometriosis patients, specifically parameters associated with the estrobolome.

DETAILED DESCRIPTION:
Patients will be recruited among the outpatient population of the National Center for Endometriosis, Department of Gynecological Surgery and Urology, Gynecology Department, University Hospital Center Zagreb following the inclusion and exclusion criteria.

To participate in the study all patients will be required to sign the Informed Consent form.

All patients will undergo a complete anamnesis via a digital form to investigate their lifestyle (occupation, stress, diet, physical activity level).

The study period will be 6 months: eight weeks on either option (verum/placebo), with an eight week washout period in between. The purpose of the washout period is to allow the gut microbiome to return to baseline. The washout period was determined based on previous gut microbiota studies with a similar design (reference), based on the fact that the gut microbiota can change rapidly (< 7 days) r.

The outcome measures (gut microbiome, quality of life) will be assessed in four distinct time points in context of the planned intervention.

T1 - before the intervention (start-of-study)

T2 - after the first intervention cycle/phase 1 (verum/placebo) of two months

T3 - after the wash-out phase of two months

T4 - after the second intervention cycle/phase 2 (verum/placebo) of two months (end-of-study)

Stool sampling will be performed with the aid of specific kits indepently by the patients. Lifestyle and quality of life will be evaluated by an online form designed specifically for the purpose of this study in Microsoft Office Forms (Microsoft, San Francisco, USA), short Online Form.

Through the process of randomization, patients will be allocated to either first receive the verum (probiotic) or the placebo (maltodextrin), and second the placebo or verum inversely.

Both patients and researchers involved will be blinded (double-blind study), the patients will be informed that they are going to take a probiotic twice for two months with a two-month time division. The intervention will consist of treatment with a multistrain probiotic formulation (Omni Biotic Stress) and the placebo which is identical in all its characteristics and packaging. Patients will be instructed to consume one sachet a day of each (probiotic) for 8 weeks and to report any symptoms or side effects related to its use. Adherence control will be carried out through the patient's notes on a separate online form provided, and also by checking the number of sachets used.

Since this is a cross-over study, data will be compared between time-points T1 and T2, and time-points T3 and T4, with the goal of minimizing the potential effect if we find that the effect of the probiotics lasted longer than eight weeks in those randomized into the intervention arm first.

ELIGIBILITY:
Minimum Age: - Maximum Age: 35 Years Sex: Female Gender Based: Ye - only women can participate in this study Accepts Healthy Volunteers: No

Inclusion Criteria:

* adult subjects with stage III or IV endometriosis diagnosis confirmed by biopsy

Exclusion Criteria:

* Age > 35 years
* Immunocompromised patients
* Patients with chronic inflammatory diseases (e.g., autoimmune disorders)
* Pregnancy
* Use of supplements and foods with probiotics
* Use of immunosuppressant, antibiotic, proton pump inhibitors and corticosteroid drugs
* Use of probiotics product less than one month before start of study or during study

Max Age: 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — just women can participate in this study
Enrollment: 40 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-05-01 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Change in relative abundance of gut microbial taxa and functional pathways related to the estrobolome in fecal samples | At baseline, after 8 weeks (end of phase 1), and after 24 weeks (end of phase 2)
  The primary outcome is the modulation of the gut microbiome. The fecal microbiome, as a genuine proxy of the gut microbiome, will be analyzed. Specific attention will be brought to taxa and metabolic pathways involved in the estrobolome.

SECONDARY OUTCOMES:
Change in quality of life measured by EHP-5 questionnaire | Week 1, Week 8, Week 16, Week 24 (6 months)
  Quality of life will be assessed using the Endometriosis Health Profile-5 (EHP-5) questionnaire at baseline, after each intervention phase, and at the end of the study.
Change in quality of life measured by SEQOL questionnaire | Week 1, Week 8, Week 16, Week 24 (6 months)
  Quality of life will be assessed using the Stellenbosch Endometriosis Quality of Life (SEQOL) questionnaire at baseline, after each intervention phase, and at the end of the study.

OTHER OUTCOMES:
Change in Mediterranean diet adherence (MEDAS score) | Week 1, Week 8, Week 16, Week 24 (6 months)
  Adherence to the Mediterranean diet will be assessed using a validated Mediterranean Diet Adherence Screener (MEDAS) at baseline and after each intervention phase
Change in perceived stress levels (PSS score) | Week 1, Week 8, Week 16, Week 24 (6 months)
  Perceived stress will be measured using the Perceived Stress Scale (PSS) questionnaire at baseline and after each intervention phase.
Change in sleep quantity (self-reported hours of sleep per night) | Week 1, Week 8, Week 16, Week 24 (6 months)
  Participants will self-report average hours of sleep per night using a standardized sleep questionnaire at baseline and after each intervention phase.
Change in physical activity levels (IPAQ score) | Week 1, Week 8, Week 16, Week 24 (6 months)
  Physical activity will be assessed using the International Physical Activity Questionnaire (IPAQ) at baseline and after each intervention phase.

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Center Zagreb, Zagreb, Croatia

IPD SHARING:
Plan to Share IPD: Undecided
That has to be decided more with the whole team